CLINICAL TRIAL: NCT07323862
Title: Spatially Transparent Binaural Beamforming for Noise Reduction for Cochlear Implant Processors
Brief Title: Assessment of a Method to Improve Cochlear Implant Users' Speech Perception in Noisy Environments While Maintaining Their Ability to Determine Where a Sound Originates From
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Vortant Technologies, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-0736; 1R43DC023172-01 (NIH)
Record Dates: First submitted 2026-01-06; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Cochlear Implant Users
Keywords: Beamforming; Speech perception in noise; Localization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Speech perception and localization with different beamformers (Experimental): Participants will listen to stimuli processed by different beamformer algorithms and repeat speech presented in noise and identify the location that sound originated from.
  Interventions: Device: Modifying audio input for cochlear implant processor

INTERVENTIONS:
Device: Modifying audio input for cochlear implant processor — Sound will be preprocessed with different beamformer algorithms and presented either through the auxiliary input port or via a streaming device to the participants' cochlear implant processor

SUMMARY:
The goal of this clinical trial is to determine if a new algorithm can improve speech perception for cochlear implant users. The main questions it aims to answer [is/are]:

* Does the algorithm improve speech perception in noisy environments?
* Does the algorithm allow listeners to determine where a sound is coming from?

Participants will

* Listen to and repeat sentences presented in the presence of noise
* Indicate the location that sounds originated from

ELIGIBILITY:
Inclusion Criteria:

* Participants must have bilateral cochlear implants from Cochlear or Advanced Bionics

Exclusion Criteria:

* Non-native English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percent correct scores on speech perception in noise. | Enrollment to 9 months
  The speech perception in noise test consists of lists of sentences in the presence of multi-talker babble or diffuse noise. The target location will vary across conditions. Participants will need to repeat back as much of the target sentence as they can.
Root mean square error for sound source localization | Enrollment to 9 months
  The localization test will involve a target speaker in the presence of multi-speaker babble or diffuse noise. The virtual location of the sound sources will be manipulated and participants will need to indicate the location of the target speaker.

CONTACTS AND LOCATIONS:
Locations (1):
- Speech and Hearing Science Building, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified behavioral IPD from all experiments will be shared with the exception of pilot data.
Time Frame: The data that will be shared will be made available no later than the time of an associated publication or one year after the end of the performance period.
  Per the policies of the Illinois Data Bank, data will be available for at least five years after it is first shared.
Access Criteria: Data that will be shared will be stored in the Illinois Data Bank, a data repository managed by the University of Illinois. The data will be publicly available via the Illinois Data Bank.